CLINICAL TRIAL: NCT02499029
Title: Glial Regulators for Treating Comorbid Posttraumatic Stress and Substance Abuse Disorders
Brief Title: N-acetylcysteine in the Treatment of PTSD and Addiction
Acronym: NAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00021986
Record Dates: First submitted 2015-07-01; First posted 2015-07-15 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: PTSD; Addiction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavior, Addictive | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetylcysteine (Experimental): Eligible participants were randomized to either NAC (2400 mg/day) or placebo for 8 weeks. The starting dose of NAC was 1200 mg twice daily (2400 mg/day). All NAC and placebo capsules contained riboflavin 25 mg, which was used as a biomarker for medication compliance.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Identical appearing placebo capsules were dispensed. All NAC and placebo capsules contained riboflavin 25 mg, which was used as a biomarker for medication compliance. Study medications (USP-grade NAC and matched placebo capsules) dispensed to participants by the medical clinician or study staff. Treatment assignment followed a pre-arranged randomization scheme and was carried out by study personnel at the pharmacy (i.e., personnel not involved in clinical management of participants to preserve the double-blind design).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — NAC pills were administered each week. NAC is a N acetyl pro-drug of the naturally-occurring amino acid cystine. NAC is a white, crystalline powder with the molecular formula C5H9NO3S and with a molecular weight of 163.2.
  Other Names: NAC
  Arms: N-Acetylcysteine
Drug: Placebo — Identical looking placebo pills were administered each week.
  Arms: Placebo

SUMMARY:
Examine the effects of N-acetylcysteine on PTSD symptoms, craving and substance use in veterans with PTSD and comorbid substance use disorders.

DETAILED DESCRIPTION:
With the increased number of military veterans returning from conflicts in Afghanistan and Iraq diagnosed with posttraumatic stress disorder (PTSD), there is a high vulnerability of these individuals to develop a substance use disorder (SUD). While there have been a host of studies focused largely on dopaminergic mechanisms of drug reward, they have not led to the development of adequate treatments for either preventing people diagnosed with PTSD from developing SUD or for treating comorbid PTSD/SUD. Based on extensive work with addictive drugs and preliminary data from our group, the investigators propose that stress impairs prefrontal cortex regulation of the basal ganglia habit circuitry and this pathology renders PTSD patients susceptible to developing SUD. Moreover, the known effects of addictive drugs to further impair prefrontal regulation are synergistic with this pathology, thereby making treatment of comorbid PTSD/SUD particularly difficult. Preclinical studies have revealed that glutamate levels within the nucleus accumbens have been implicated in drug seeking behavior in the animal model of relapse. The amino acid precursor N-acetylcysteine (NAC) appears to restore glutamate to normal levels and may also prevent glutamate levels from spiking following subsequent stimulant use. The primary goal of the proposed study is to evaluate the efficacy and safety of N-acetylcysteine in preventing relapse in drug dependent individuals with PTSD or subthreshold PTSD. Veterans with substance use disorders who have achieved at lease one week of abstinence will be randomized to either placebo or NAC (2400-3600mg/day) for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old
* U.S. military Veteran, Reservist, or National Guard member
* DSM-IV diagnostic criteria for current (past 6 months) SUD and PTSD or subthreshold PTSD (i.e., met criteria for cluster B (re-experiencing) and either cluster C (avoidance) or D (hyperarousal), as well as duration of one month and clinically significant impairment)
* Score of > 21 on the Mini-Mental State Exam (MMSE).

Exclusion Criteria:

* Unstable medical conditions
* Bipolar or psychotic disorders
* Seizures or asthma
* Prior treatment with NAC
* Suicidality
* Enrolled in ongoing PTSD treatment (pharmacotherapy or psychosocial)
* Females: could not be pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

REFERENCES:
- [Result] Back SE, McCauley JL, Korte KJ, Gros DF, Leavitt V, Gray KM, Hamner MB, DeSantis SM, Malcolm R, Brady KT, Kalivas PW. A Double-Blind, Randomized, Controlled Pilot Trial of N-Acetylcysteine in Veterans With Posttraumatic Stress Disorder and Substance Use Disorders. J Clin Psychiatry. 2016 Nov;77(11):e1439-e1446. doi: 10.4088/JCP.15m10239. PMID 27736051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the VA medical center between March 2013 and April 2014.
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 18 | 17
Completed | 13 | 14
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (8.6) | 49.9 (8.1) | 49.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 27
Substance Use Disorder (SUD) [Count of Participants; unit: Participants]
  Alcohol | 10 | 12 | 22
  Cocaine | 11 | 9 | 20
  Opioid | 0 | 1 | 1
Post Traumatic Stress Disorder (PTSD) [Mean (Standard Deviation); unit: units on a scale] — PTSD was measured using the CAPS IV and the PCL-M.
  The CAPS IV measures seventeen symptoms based on intensity and frequency. Intensity and frequency scores are summed to create a severity score. Severity scores are summed to get a total score. A higher total score indicates a higher severity of PTSD symptoms. The full range for CAPS IV is 0-136.
  The PCL-M is a seventeen question self-report, scored on a scale from 1 to 5, with possible scores from 17 to 85. The scores are summed to get a total score. A higher total indicates a higher severity of PTSD symptoms.
  units on a scale
    CAPS IV | 58.8 (21.2) | 68.6 (23.7) | 63.8 (22.6)
    PCL-M | 45.7 (14.6) | 43.4 (18.6) | 44.5 (16.5)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: Clinician Administered PTSD Scale IV (CAPS) The CAPS IV measures seventeen symptoms based on intensity and frequency. Intensity and frequency scores are summed to create a severity score for each question. Severity scores are summed to get a total score. A higher total score indicates a higher severity of PTSD symptoms.The full range for CAPS IV is 0-136.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale
  4 Weeks | 38.7 (20.0) | 52.8 (36.9)
  8 Weeks | 32.0 (23.5) | 51.5 (43.1)

2. Secondary Outcome: Depression
Description: Beck Depression Inventory (BDI) The BDI measures presence and severity of depression. It has 21 questions that are rated from 0-3 with a highest possible score of 63. A higher score indicates a higher severity of depression.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale
  Week 4 | 10.9 (6.4) | 18.5 (14.8)
  Week 8 | 9.9 (6.7) | 19.3 (15.8)

3. Secondary Outcome: Craving
Description: Visual Analogue Scale (VAS) The VAS measures alcohol craving on a scale from 0 to 10. A higher score indicates a higher level of craving.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale
  Amount of Craving Week 4 | 1.8 (1.9) | 2.8 (2.6)
  Amount of Craving Week 8 | .7 (.7) | 2.8 (2.8)
  Frequency of Craving Week 4 | 1.8 (2.0) | 2.4 (2.3)
  Frequency of Craving Week 8 | 1.0 (.9) | 3.0 (2.9)
  Intensity of Craving Week 4 | 1.8 (2.1) | 2.9 (2.8)
  Intensity of Craving Week 8 | 1.3 (1.9) | 2.8 (3.1)

4. Secondary Outcome: PTSD Symptoms
Description: PTSD Checklist - Military (PCL-M) The PCL-M is a seventeen question self-report, scored on a scale from 1 to 5, with possible scores ranging from 17 to 85. The scores from each question are summed to get a total score (17-85). A higher total indicates a higher severity of PTSD symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale
  Week 4 | 33.8 (10.6) | 41.9 (21.7)
  Week 8 | 31.2 (9.7) | 41.9 (22.8)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; A series of hierarchical linear regression analyses were conducted to examine the effects of treatment group (NAC or placebo) on PTSD symptomatology, craving, substance use, and depression. Baseline levels of the respective outcome measures were entered in Step 1 of the model to adjust for any baseline differences. Treatment group was entered as the predictor in Step 2. The significance threshold was set at a p-value of .05 (two-sided) for all statistical tests; Test type: Superiority; p = .05, Regression, Linear

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/17
Other Adverse Events (participants affected / at risk) | 12/18 | 7/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetylcysteine (N=18) | Placebo (N=17)
Cardiac Arrhythmia (Cardiac disorders) | 1 | 0
Syncopal Episode (Blood and lymphatic system disorders) | 0 | 1
Suicidality (Psychiatric disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Death (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetylcysteine (N=18) | Placebo (N=17)
Dry Mouth (General disorders) | 0 | 2
Abdominal Burning (Gastrointestinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (General disorders) | 0 | 1
Fungal Rash (Infections and infestations) | 0 | 1
Heartburn (Gastrointestinal disorders) | 2 | 0
Hot Flashes (General disorders) | 1 | 0
Mood Changes (Psychiatric disorders) | 0 | 1
Poison Oak Rash (Infections and infestations) | 1 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tingling Left Arm (General disorders) | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 0 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Spider Bite (Infections and infestations) | 1 | 0
Unstable Cardiac Condition (Cardiac disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small sample size, Veterans only which may limit ability to generalize to other populations, self-report measures may introduce bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No